CLINICAL TRIAL: NCT05109481
Title: EVALUATION OF IMPACT OF THE MASK ON THE VISUAL PREFERENCES OF THE NEWBORN
Brief Title: Masks and Visual Preferences in the Newborn
Acronym: BABYMASK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01711-40
Record Dates: First submitted 2021-09-22; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-09

CONDITIONS: Newborn; Vision, Ocular; Masks
Keywords: Neonatology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What impact can facial masks have on face exploration in the first few weeks of life? No study has yet investigated this. The objective of our study was to evaluate the impact of the mask on the face processing (preferential gaze, visual recognition) of the term infant for familiar (e.g. mother's face) and unfamiliar (stranger's face) faces.

This is a prospective study which will take place in Grenoble Maternity Hospital.

200 newborns will be enrolled between 24 hours and 7 days of life during one year. Different pairs of images will be presented on a screen while an experimenter records the infant's gaze. On each trial, the experimenter will judge when the infant is looking at the screen or not and assess when 10 seconds of screen gaze time has been accumulated.

The comparisons will be made to determine whether statistically, one face is looked at significantly longer than another.

DETAILED DESCRIPTION:
Background Since March 2020, the mask has invaded the everyday life of families, workplaces and hospitals. In contrast to the pre-Covid era, healthy newborns in their first days of life are now exposed to the faces of adults wearing masks. Yet early visual experience of newborns with faces is crucial, as it will set the stage for early communication .For example, a systematic preference for human faces exists in newborns .However, this system is not limited to a preferential orientation; it has been shown that the newborn recognises faces during the first week of life .

Maternal recognition is particularly important for the development of attachment and emotional interactions. Several studies have shown that 2-3 day old infants recognize their mother's face (real, in vivo) despite relatively limited visual acuity .However, no study has been able to show the same on the basis of photographs (without other sensory stimuli), such as the mother's smell.

Objective The aim of this study is to measure the impact that these masks can have on the exploration of known (mother) and unknown faces in the first weeks of life. No study has so far investigated this.

Methods Study This is a prospective, single-centre study.

Population The newborns included will be newborns between 24 hours and 7 days of life before discharge from the maternity hospital, born at term (37 weeks of gestational age) at the Grenoble University Hospital, whose parents speak French, are beneficiaries of social security, and did not object to participating in the study. Newborns with a pathology requiring or having required examinations, hospitalisation or other during the first 24 hours, which could have impacted on the exposure of the newborn to the mask or parents suffering from Covid during the maternity stay will not be included in the study.

Protocol For a newborn, each test will take place between 24 hours and discharge from the maternity hospital (generally <7 days) for a newborn. Concerning the test: the newborns are installed on the mother's, facing the computer screen above which is positioned the experimenter in charge of recording the infants' gaze. The screen is positioned 30 cm from the newborns' face, a distance appropriate to their poor visual acuity.

The investigators are going to carry out visual preference tests. This involves pairs of images presented on the screen while an experimenter records the infant's gaze. On each trial, the experimenter will judge when the infant is looking at the screen or not and assess when 10 seconds of screen time has been accumulated.

Ideally, a newborn should be able to do a series of trials, but as their attention fluctuates according to the time of day and from one individual to another, it is possible that some children may only do one trial.

Statistical analysis A minimum of 30 participants per test will be required. As not all infants tested can be included in our study, because they are likely to fall asleep, become restless or exhibit maladaptive behaviour (approximately 30%), the invetigators will test 200 children for the 5 tests. The behavioural data consist of gaze times on stimuli during a presentation period. The behavioural data consist of gaze times on stimuli during a presentation period. These gaze times are obtained by manually scanning the videos. Comparisons of the mean of the proportions of gaze times to each image will be made with parametric tests (Student's t test, analysis of variance or mixed models if n = 30 in each test) or non-parametric tests (Chi-2, if n < 30 in each group) in order to determine whether statistically, one face is gazed at significantly longer than another. Using Gpower software, a moderate effect size was estimated for a sample of 20 newborns (estimated statistical power of 0.8).

Expected results Our hypothesis and clinical impression is that the mask has an impact on the visual exploration of the neonate. The investigators expect that the effects will also be modulated by the neonate's visual experience with the mask but also by the information requested in the "mask exposition" questionnaire. Indeed, these characteristics may influence the newborn's experience with masked and unmasked faces, as well as the quality of mother-infant interactions.

ELIGIBILITY:
Inclusion Criteria:

* newborns between 24 hours and 7 days of life before discharge from the maternity hospital,
* born at term (37 weeks of gestational age) at the Grenoble University Hospital,
* whose parents speak French
* whose parents are beneficiaries of social security
* whose parents did not object to participating in the study.

Exclusion Criteria:

Newborns with

* a pathology requiring or having required examinations,
* a hospitalisation or other during the first 24 hours, which could have impacted on the exposure of the newborn to the mask
* parents suffering from Covid during the maternity stay will not be included in the study.

Ages: 24 Hours to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 200 healthy newborn born between September 2021 ans September 2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Time of fixation of the newborn's gaze on an image | One year
  Time of fixation of the newborn's gaze on an image

IPD SHARING:
Plan to Share IPD: No